CLINICAL TRIAL: NCT00214331
Title: Pharmacokinetics and Pharmacodynamics and Selected Antibiotics During Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2002-524; FDA # 233-02-0114
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy
MeSH Terms: interventions — Ciprofloxacin; Azithromycin; Gentamicins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: ciprofloxacin
  Interventions: Drug: ciprofloxacin
- 2: azithromycin
  Interventions: Drug: azithromycin
- 3: gentamicin
  Interventions: Drug: gentamicin

INTERVENTIONS:
Drug: ciprofloxacin — ciprofloxacin 500 mg twice a day for five doses.
  Groups: 1
Drug: azithromycin — azithromycin 500 mg on day 1 followed by 250 mg on days 2-5
  Groups: 2
Drug: gentamicin — a single intravenous dose of gentamicin 1.5mg/kg infused over 60 minutes
  Groups: 3

SUMMARY:
This protocol is a prospective, open-label, multicenter, population pharmacokinetic and pharmacodynamic study of selected anti-infective agents in pregnant women being treated for suspected or documented infections.

ELIGIBILITY:
Inclusion Criteria:

* Women in their second or third trimester of pregnancy
* Women currently receiving treatment or whose physician has made the decision to start treatment with ciprofloxacin, azithromycin or gentamicin for a suspected or documented infection
* Of childbearing potential and who either have never been pregnant or whose most recent pregnancy ended 3 months previously (control group)
* Women greater than 3 months postpartum and currently breast-feeding (substudy)

Exclusion Criteria:

* Women with significant gastrointestinal disease which may be expected to interfere with the absorption of the orally administered anti-infective agents

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who are prescribed antibiotics as part of their clinical care
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2003-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Sarto, MD, PhD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States